CLINICAL TRIAL: NCT05963347
Title: A Phase 2 Study to Investigate the Safety, Tolerability and Anti-tumor Activity of Golidocitinib in Combination With CHOP as the Front-line Treatment for Participants With Peripheral T-cell Lymphomas (PTCL)
Brief Title: Go-CHOP as the Frontline Therapy for PTCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, KeshuZhou, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022J0003
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Go-CHOP (Experimental): Golidocitinib in combination with CHOP
  Interventions: Drug: Golidocitinib; Drug: CHOP Regimen

INTERVENTIONS:
Drug: Golidocitinib — Daily dose. Starting dose of golidocitinib is 75 mg QD. If tolerated, subsequent cohorts will test ascending doses of golidocitinib.
  Other Names: AZD4205, DZD4205
Drug: CHOP Regimen — CHOP will be administered in a 21-day cycle for a maximum of 6 cycles.
  Other Names: Cyclophosphamide, doxorubicin, vincristine, prednisone

SUMMARY:
This is a phase 2 Study to investigate the safety, tolerability, and anti-tumor activity of golidocitinib in Combination with CHOP as the front-line Treatment for Participants with Peripheral T-cell Lymphomas (PTCL).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign an informed consent form prior to trial-specific procedures, sampling, and analysis.
2. Participants must be at least 18 years of age (inclusive) at the time of signing the informed consent form.
3. The participant has an ECOG performance status of 0 to 2 and has not deteriorated in the past 2 weeks.
4. Life expectancy ≥ 3 months.
5. Histologically confirmed diagnosis of PTCL and no prior systemic anti-lymphoma therapy; and assessed by a local pathologist according to the 2016 revised World Health Organization Classification of Lymphoid Tumors (Swerdlow SH et al., 2017) as the following subtypes:

   * peripheral T-cell lymphoma, not otherwise specified (PTCL, NOS)
   * angioimmunoblastic T cell lymphoma (AITL)
   * follicular T-cell lymphoma (FTCL)
   * nodular PTCL with follicular helper T-cell phenotype (nodular PTCL with TFH phenotype)
   * ALK- anaplastic large cell lymphoma (ALK- ALCL)
   * ALK+ anaplastic large cell lymphoma (ALK + ALCL)
   * enteropathy-associated T-cell lymphoma (EATL)
   * monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL)
   * hepatosplenic T-cell lymphoma (HSTCL)
   * subcutaneous panniculitis-like T-cell lymphoma (SPTCL)
6. Adequate bone marrow reserve and organ system function reserve
7. Left ventricular ejection fraction (LVEF) ≥ 50% as assessed by ECHO.
8. Participants should be able and willing to comply with the study protocol requirement.
9. Adequate birth control measures should be taken during study treatment and the corresponding washout period.

Exclusion Criteria:

1. Received any of the following interventions:

   * Prior therapy for PTCL prior to enrollment, except short-term corticosteroids (duration ≤ 7 days, equivalent prednisone dose ≤ 15 mg/day).
   * Prior radiation therapy for PTCL except local therapy for individual areas.
   * Currently receiving other systemic antineoplastic or investigational therapy.
   * Participants who have received more than 200 mg/m2 doxorubicin or other equivalent doses of anthracycline/anthraquinone (e.g., epirubicin, daunorubicin, mitoxantrone, etc.) cumulatively.
   * Major surgical procedures (excluding routine lymphoma care programs such as vascular access placement, biopsy, etc.) or significant trauma within 4 weeks prior to the first dose of study treatment, or anticipation of the need for major surgery during the study.
   * Prior treatment with JAK or STAT3 inhibitors following diagnosis of PTCL.
   * Live vaccine within 28 days prior to enrollment.
   * Participants currently receiving (or unable to discontinue for at least 1 week prior to first dose) vitamin K antagonists, antiplatelets, or anticoagulants.
   * Participants currently receiving (or unable to discontinue for at least 1 week prior to receiving the first dose) medications or herbal supplements known to be highly potent inhibitors or inducers of CYP3A or sensitive substrates of BCRP or P-gp with a narrow therapeutic index (see Section 6.8).
2. Participants with clinical manifestations or imaging findings suggesting central nervous system or leptomeningeal lymphoma.
3. Participants with severe lung dysfunction, pneumonitis, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, or any prior history of clinically active interstitial lung disease.
4. Participants with a condition that requires treatment with immunosuppressants, biologics, or nonsteroidal anti-inflammatory drugs (NSAIDs).
5. Participants with active infections
6. Participants with significant cardiac disorder
7. Other malignancies within 3 years before enrollment. However, malignancies, such as uterine and cervical carcinoma in situ, basal or squamous cell carcinoma, and non-melanotic skin cancer, which have been clinically cured after evaluation, may be considered for inclusion after evaluation.
8. Refractory nausea or vomiting that cannot be controlled by supportive therapy, chronic gastrointestinal disease, inability to swallow pharmaceutical agents or previous major bowel resection may affect the adequate absorption of golidocitinib.
9. Female participants who are lactating.
10. Participants with a history of hypersensitivity against the active ingredients or excipients of golidocitinib or against similar chemical structures or drugs of the same class. Contraindication to any agent in the CHOP chemotherapy regimen.
11. Participants with any severe or poorly controlled systemic disease, such as poorly controlled hypertension or active bleeding constitution, as judged by the investigator or other evidence.
12. Participants with an intercurrent illness that, in the opinion of the investigator, may jeopardize compliance with the protocol, including any significant medical condition, laboratory abnormality, or psychiatric disorder.
13. Participants with psychological, familial, social, or geographical conditions that preclude compliance with the program. Any condition that would confound the ability to interpret study data.
14. Participating in study planning and implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From first dose till 28 days post the last dose
  TEAE, lab test

SECONDARY OUTCOMES:
Complete Response Rate | From date of enrollment (first dose) until the end of induction therapy completed (~ 18 weeks)
  Complete response rate by Cycle 3 and Cycle 6 assessed by investigator per Lugano 2014 criteria
Objective Response Rate | From date of enrollment (first dose) until the end of induction therapy completed (~ 18 weeks)
  Objective response rate by Cycle 3 and Cycle 6 assessed by investigator per Lugano 2014 criteria.
Progression Free Survival | From date of enrollment (first dose) until documented disease progression or death of any reason (up 2 year)
  Objective response rate by Cycle 3 and Cycle 6 assessed by investigator per Lugano 2014 criteria.
Duration of Response | from first documented response till disease progression or death of any reason (up to 2 years)
  Duration of response assessed by investigator per Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Keshu Zhou, Dr., Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No